CLINICAL TRIAL: NCT01602172
Title: Trial of Nurse-delivered Alcohol Brief Intervention for Hospitalized Veterans
Brief Title: Health Behavior Change for Hospitalized Veterans
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitment challenges. Extensive remedial recruitment strategies unsuccessful
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: NRI 11-339
Record Dates: First submitted 2012-05-16; First posted 2012-05-18 (Estimated); Results first posted 2019-09-09 (Actual); Last update posted 2019-09-17 (Actual); Status verified 2019-09

CONDITIONS: Alcohol Consumption
Keywords: alcohol consumption; inpatients; risk reduction behavior; counseling; nurses; brief intervention
MeSH Terms: conditions — Alcohol Drinking; Risk Reduction Behavior | interventions — Ethanol; Methods

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Brief Alcohol Intervention (BI) (Experimental): The 3-part Brief Intervention (BI) consists of . Part I is 15-minute multi-component motivational discussion in hospital which includes personalized risk feedback, advice to abstain or reduce consumption, and the negotiation of an individual change plan. Part II is 15-minute follow-up in hospital to reinforce Part I. Part III is 15-minute follow-up telephone call at 2 weeks to reinforce Part I.
  Interventions: Behavioral: Brief Alcohol Intervention
- Attention Control (Active Comparator): These subjects receive a set of Lifestyle brochures which contain information and tips for healthy lifestyle behaviors such as alcohol and tobacco use, weight management, and physical activity. Two weeks later, the Research Assistant calls subjects in this condition at home for a 5-15 minute session to review the brochures and discuss any questions that s(he) may have. This intervention is designed to provide all the information and assessments that that Brief Intervention participants as well as all the alcohol consumption and motivation to change measures-- it is designed to control for the attention that the BI participants receive w/o the motivational interventions
  Interventions: Other: Lifestyle brochures
- Control (Active Comparator): These subjects receive a set of Lifestyle brochures which contain information and tips for healthy lifestyle behaviors such as alcohol and tobacco use, weight management, and physical activity to discuss with the Research Assistant. Approximately two weeks later, the Research Assistant will call patients in this condition at home for a 5-15 minute session to review the brochures and discuss any questions that s(he) may have. Subjects complete only drinking quantity measures at baseline and 6 months post baseline. The inclusion of this group tests whether completing more extensive questionnaires (in comparison the Attention Control group) decreases alcohol consumption.
  Interventions: Other: Lifestyle brochures

INTERVENTIONS:
Behavioral: Brief Alcohol Intervention — 3 part intervention: Part I is 15-minute multi-component motivational discussion in hospital which includes personalized risk feedback, advice to abstain or reduce consumption, and the negotiation of an individual change plan. Part II is 15-minute follow-up in hospital to reinforce Part I. Part III is 15-minute follow-up telephone call at 2 weeks to reinforce Part I.
  Arms: Brief Alcohol Intervention (BI)
Other: Lifestyle brochures — Set of educational brochures/brochures which contain information and tips for healthy lifestyle behaviors such as alcohol and tobacco use, weight management, and physical activity to discuss with the Research Assistant. Approximately two weeks later, the Research Assistant will call patients in this condition at home for a 5-15 minute session to review the brochures and discuss any questions that s(he) may have.
  Arms: Attention Control; Control

SUMMARY:
Veterans drink, binge drink, and drive under the influence of alcohol at higher rates than non-Veterans do. Addressing alcohol misuse, the range of alcohol consumption from risky drinking to alcohol abuse and alcoholism, is a national priority for the VA. It is recommended that people keep their alcohol consumption below limits established by the National Institutes of Health (NIH). A type of 10-15 minute counseling known as "brief intervention" (BI) has been shown to help risky drinkers cut back to the NIH-recommended limits. This study will examine the impact of a nurse-delivered alcohol BI on hospitalized Veterans' weekly number of drinks, monthly number of binge drinking episodes, readiness to change drinking behavior, and alcohol-related problems. This preventative approach for reducing alcohol consumption is intended to help Veterans avoid many of the physical and psychosocial consequences of alcohol misuse.

DETAILED DESCRIPTION:
Improving the identification and management of alcohol misuse is a VA priority. Alcohol misuse includes the spectrum of alcohol consumption ranging from hazardous drinking to alcohol use disorders (alcohol abuse and dependence). The VA recommends using a set of clinical strategies referred to as Screening, Brief Intervention, and Referral to Treatment (SBIRT) to identify and address alcohol misuse in primary care settings. Brief intervention (BI), a core component of SBIRT, significantly reduces alcohol consumption, morbidity, and healthcare utilization in hazardous drinkers, but its efficacy is not well-established outside of outpatient settings. In the hospital setting, nurses are well-positioned to deliver BI, but research is needed to determine the efficacy of inpatient nurse-delivered BI, particularly with hazardous drinkers. The few previous trials of BI in the inpatient setting demonstrated limited effects on alcohol consumption and alcohol-related problems, potentially due to assessment reactivity--extensive patient assessment that inadvertently raises patient awareness about drinking in both groups, mimicking the effect of BI and thus driving findings towards the null. Additionally, very few of these trials involved nurse delivery of the intervention and many included patients with alcohol use disorders, patients believed to be beyond the "therapeutic reach" of BI.

The primary goal of this 3-arm randomized controlled trial is to examine the efficacy of nurse-delivered alcohol BI with hospitalized patients who are hazardous drinkers and to identify barriers and facilitators to implementation of BI in inpatient settings. Arm 1 (BI) consists of Veterans randomized to nurse-delivered BI, Arm 2 (AC) consists of Veterans randomized to an attention control, and Arm 3 (AC-LA) consists of Veterans randomized to an attention control with limited assessment of readiness to change and adverse consequences of alcohol use so as to reduce and evaluate assessment reactivity.

Specific Aim 1 is to determine the impact of a nurse-led BI on the alcohol screening status, number of drinks/week, number of binge drinking episodes, readiness to change drinking behavior, and adverse consequences of alcohol use in hospitalized hazardous drinkers. Specific Aim 2 is to formatively evaluate the process of the intervention implementation to inform the design and execution of a future, multi-site randomized effectiveness trial of the intervention. A secondary aim is to identify factors, issues, and themes related to Veterans' interest and motivation for changing their alcohol consumption.

We will recruit 320 hospitalized Veterans admitted to one of the three medical-surgical units at the VA Pittsburgh Healthcare System. Veterans will be included who are >21 years old, able to speak English, and are hazardous, non-dependent drinkers, as defined by criteria established by the National Institute for Alcohol Abuse and Alcoholism and by the Composite International Diagnostic Interview Substance Abuse Module. Patients randomized to Arm 1 will receive a three-part nurse-delivered BI. Patients randomized to Arms 2 and 3 will receive usual care plus healthy lifestyle brochures addressing general healthy lifestyle behaviors, such as limited alcohol consumption, tobacco cessation, and weight management. For Specific Aim 1, we will use various multivariable linear and logistic regressions that account for continuous outcomes, dichotomous outcomes, and clustering within medical units. Poisson regressions or negative binomial regressions will be used if the continuous outcome measures are not normally distributed. For Specific Aim 2, we will use basic descriptive statistics in order to describe the numbers of deviations and interruptions to intervention delivery as planned. Based on interventionist field notes, we will categorize the types of deviations/interruptions. We will also use these descriptive statistics to describe duration of the audio-recorded intervention; the presence/absence of various techniques within the BI; the receipt/nonreceipt of additional alcohol feedback, advice, or counseling; and patient responsiveness to/perceptions of the BI. We will also code brief free-text perceptions responses using a modified grounded theory approach.

ELIGIBILITY:
Inclusion Criteria:

* U.S. Veterans admitted to one of the three medical-surgical units at VA Pittsburgh Healthcare System (VAPHS)
* age 21 years or older
* ability to speak English
* hazardous, non-dependent alcohol consumption

Exclusion Criteria:

* Alcohol dependence (as determined using Section C (Alcohol) from the Composite International Diagnostic Interview Substance Abuse Module (CIDI-SAM)
* Current participation (past 6 months) in substance abuse treatment or 12-step program
* age <21 years
* significant cognitive impairment (as determined by the Short Blessed test , score >10)
* bipolar disorder or active psychosis
* sensory impairment precluding communication
* medically-related inability to participate or consent to study participation
* current pregnancy
* current incarceration
* lack of telephone access or unwillingness to be contacted for follow-up
* enrollment in the study during a prior inpatient admission at VAPHS
* current enrollment in other substance use trials (due to the potential influence of dual participation on study outcomes)

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2012-12; Primary Completion 2015-01 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lauren M. Broyles, PhD RN, Principal Investigator — VA Pittsburgh Healthcare System University Drive Division, Pittsburgh, PA
Locations (1):
- VA Pittsburgh Healthcare System University Drive Division, Pittsburgh, PA, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Broyles LM, Wieland ME, Confer AL, Youk AO, Gordon AJ. Holes in the pipeline: addressing recruitment challenges for an alcohol brief intervention trial in the acute care setting. [Abstract]. Substance Abuse. 2014 Jan 1; 35(2):208.
- [Result] Broyles LM, Wieland ME, Confer AL, DiNardo MM, Kraemer KL, Hanusa BH, Youk AO, Gordon AJ, Sevick MA. Alcohol brief intervention for hospitalized veterans with hazardous drinking: protocol for a 3-arm randomized controlled efficacy trial. Addict Sci Clin Pract. 2015 May 13;10(1):13. doi: 10.1186/s13722-015-0033-6. PMID 25968121
- See also: Recruitment is described in full in this open access article. — http://www.ascpjournal.org/content/pdf/s13722-015-0033-6.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment occurred December 2012 to June 2014 on three medical-surgical units at the VA Pittsburgh Healthcare System.
Pre-assignment Details: Not applicable; no enrolled participants were excluded from the trial prior to randomization.
Groups:
- Brief Alcohol Intervention (BI): Brief Intervention Condition--3 part motivational discussion in and out of hospital
  Brief Alcohol Intervention: 3 part intervention: Part I was a 15-minute multi-component motivational discussion in hospital which included personalized risk feedback, advice to abstain or reduce consumption, and the negotiation of an individual change plan. Part II was a 15-minute follow-up in hospital to reinforce Part I. Part III was 15-minute follow-up telephone call at 2 weeks to reinforce Part I.
- Attention Control: Traditional Attention Control Condition
  Lifestyle brochures: Set of educational brochures/brochures which contained information and tips for healthy lifestyle behaviors such as alcohol and tobacco use, weight management, and physical activity to discuss with the Research Assistant. Approximately two weeks later, the Research Assistant called patients in this condition at home for a 5-15 minute session to review the brochures and discuss any questions that s(he) had.
- Control: Attention Control, Limited Assessment
  Lifestyle brochures: Set of educational brochures/brochures which contained information and tips for healthy lifestyle behaviors such as alcohol and tobacco use, weight management, and physical activity to discuss with the Research Assistant. Approximately two weeks later, the Research Assistant called patients in this condition at home for a 5-15 minute session to review the brochures and discuss any questions that s(he) had.
Period: Overall Study
Arm/Group | Brief Alcohol Intervention (BI) | Attention Control | Control
Started | 37 | 23 | 22
Completed | 32 | 17 | 22
Not Completed | 5 | 6 | 0

BASELINE CHARACTERISTICS:
Groups:
- Brief Alcohol Intervention (BI): Brief Intervention Condition--3 part motivational discussion in and out of hospital
  Brief Alcohol Intervention: 3 part intervention: Part I is 15-minute multi-component motivational discussion in hospital which includes personalized risk feedback, advice to abstain or reduce consumption, and the negotiation of an individual change plan. Part II is 15-minute follow-up in hospital to reinforce Part I. Part III is 15-minute follow-up telephone call at 2 weeks to reinforce Part I.
- Attention Control: Traditional Attention Control Condition
  Lifestyle brochures: Set of educational brochures/brochures which contain information and tips for healthy lifestyle behaviors such as alcohol and tobacco use, weight management, and physical activity to discuss with the Research Assistant. Approximately two weeks later, the Research Assistant will call patients in this condition at home for a 5-15 minute session to review the brochures and discuss any questions that s(he) may have.
- Control: Attention Control, Limited Assessment
  Lifestyle brochures: Set of educational brochures/brochures which contain information and tips for healthy lifestyle behaviors such as alcohol and tobacco use, weight management, and physical activity to discuss with the Research Assistant. Approximately two weeks later, the Research Assistant will call patients in this condition at home for a 5-15 minute session to review the brochures and discuss any questions that s(he) may have.
- Total: Total of all reporting groups
Arm/Group | Brief Alcohol Intervention (BI) | Attention Control | Control | Total
Number analyzed (Participants) | 37 | 23 | 22 | 82
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.3 (13.16) | 62.70 (9.10) | 58.68 (11.02) | 59.18 (11.67)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 0 | 0 | 2
  Male | 35 | 23 | 22 | 80
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 31 | 19 | 19 | 69
  Race: Black | 6 | 4 | 3 | 13
Alcohol Use Disorders Identification Test-Consumption [Mean (Standard Deviation); unit: units on a scale] — AUDIT-C scores range from 0-12, with higher values representing a worse outcome (a score of 4 indicating hazardous drinking in males and 3 hazardous drinking in females).
  units on a scale | 6.11 (2.47) | 7.43 (2.25) | 6.36 (1.97) | 6.54 (2.33)
Weekly number of drinks [Mean (Standard Deviation); unit: count of drinks per week] | 17.36 (16.53) | 20.78 (14.76) | 18.04 (11.81) | 18.52 (14.77)
Number of Binge Episodes/Week [Mean (Standard Deviation); unit: count of binge episodes per week] | 4.22 (7.31) | 7.61 (9.90) | 5.36 (8.68) | 5.48 (8.48)
Socrates Score [Mean (Standard Deviation); unit: units on a scale] — Socrates - Taking Steps Subscale assesses readiness to change drinking behavior.
  Socrates (Stages of Change Readiness and Treatment Eagerness Scale). A 19-item instrument with 3 subscales where minimum score is 19 and the maximum is 95. Lower totals representing lesser readiness/eagerness for change. With the three sub scales (Recognition, Ambivalence, and Taking Steps), higher scores indicate greater recognition, ambivalence and taking steps and scores range from 7 to 35, 4 to 20, and 8 to 40, respectively. Population: Only participants in the two active groups completed this scale
  units on a scale
    number analyzed (Participants) | 37 | 23 | 0 | 60
    (all) | 21.86 (8.43) | 16.52 (10.48) |  | 19.82 (4.72)
SIP-2R Score [Mean (Standard Deviation); unit: units on a scale] — Short Inventory of Problems Score-2R. SIP-2R was used as a continuous measure with possible scores from 0-45, where each item has a score from 0-3 (0=Never, 1=once or a few times, 2=once or twice a week, 3=daily or almost daily). Higher scores indicate a worse outcome. Population: Only participants in the two active groups completed this scale
  units on a scale
    number analyzed (Participants) | 37 | 23 | 0 | 60
    (all) | 4.43 (5.19) | 5.17 (9.24) |  | 4.72 (6.96)

OUTCOME MEASURES:

1. Primary Outcome: Number of Standard Drinks Per Week
Description: Number of Drinks per Week was determined by the product of responses to the following two NIAAA questions during the recruitment and screening processes : (1) On average, how many days a week do you have an alcoholic drink?; (2) On a typical drinking day, how many standard-sized drinks do you have? (Appendix 2). "Standard-sized drink" will refer to 12 ounces beer, 5 ounces wine, or 1.5 ounces liquor/spirits.
Time Frame: 6 months
Population: Reflects number of participant that completed the 6 month interview
Measure: Mean (Standard Deviation); unit: days/week drink * amt of drinks in day
Groups:
- Brief Intervention: 3-part Brief Intervention
  Brief Alcohol Intervention: 3 part intervention: Part I is 15-minute multi-component motivational discussion in hospital which includes personalized risk feedback, advice to abstain or reduce consumption, and the negotiation of an individual change plan. Part II is 15-minute follow-up in hospital to reinforce Part I. Part III is 15-minute follow-up telephone call at 2 weeks to reinforce Part I.
- Control: Control, Limited Assessment
  Lifestyle brochures: Set of educational brochures/brochures which contain information and tips for healthy lifestyle behaviors such as alcohol and tobacco use, weight management, and physical activity to discuss with the Research Assistant. Approximately two weeks later, the Research Assistant will call patients in this condition at home for a 5-15 minute session to review the brochures and discuss any questions that s(he) may have.
Arm/Group | Brief Intervention | Attention Control | Control
Number analyzed (Participants) | 32 | 17 | 22
days/week drink * amt of drinks in day | 11.19 (14.39) | 13.12 (10.93) | 14.00 (4.05)

2. Secondary Outcome: Alcohol Screening Status
Description: Alcohol Screening Status will be assessed using the Alcohol Use Disorders Identification Test-Consumption (AUDIT-C) (Appendix 2), the 3-item short form of the 10-item Alcohol Use Disorders Identification Test (AUDIT) developed by the World Health Organization. AUDIT-C data will be collected during the recruitment and screening processes. AUDIT-C scores range from 0-12, with higher values representing a worse outcome (a score of 4 indicating hazardous drinking in males and 3 hazardous drinking in females).Generally, the higher the AUDIT-C score, the more likely it is that the patient's drinking is affecting his/her health and safety.
Time Frame: 6 months
Population: Only participants that completed the 6 month interview
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Brief Intervention | Attention Control | Control
Number analyzed (Participants) | 32 | 17 | 22
units on a scale | 5.09 (3.03) | 5.41 (2.98) | 5.27 (2.35)
Statistical Analysis 1: Comparison: Brief Intervention vs Attention Control vs Control; Measures were compared with linear mixed effects regression models to compare impact of BI compared to usual care conditions. Analyses reported here included only those that completed the 6 month interview (71/82 baseline participants); Test type: Equivalence — Results of the regression models were used to reject null hypotheses of equivalence with p-values of comparisons across groups in changes in alcohol related measures using p-values < 0.05 as significant; p = .05, Mixed Models Analysis — First, significance of the regression model was viewed. When the overall model was significant, tests of the co-efficients were viewed. Primary effects of interest were the treatment group X time interactions

3. Secondary Outcome: Number of Binge Drinking Episodes Over Past 30 Days
Description: Number of Binge Drinking Episodes will be assessed through a third NIAAA question during the recruitment and screening processes: (3) How many times in the past 30 days have you had 5 or more standard-sized drinks in a day (men), or 4 or more standard-sized drinks in a day? (women)
Time Frame: 6 months
Population: Participants the completed the 6 month interviews
Measure: Mean (Standard Deviation); unit: binge drinking episodes
Groups:
- Attention Control: Attention Control Condition
  Lifestyle brochures: Set of educational brochures/brochures which contain information and tips for healthy lifestyle behaviors such as alcohol and tobacco use, weight management, and physical activity to discuss with the Research Assistant. Approximately two weeks later, the Research Assistant will call patients in this condition at home for a 5-15 minute session to review the brochures and discuss any questions that s(he) may have.
Arm/Group | Brief Intervention | Attention Control | Control
Number analyzed (Participants) | 32 | 17 | 22
binge drinking episodes | 2.25 (4.72) | 4.65 (7.72) | 4.14 (8.29)

4. Secondary Outcome: Readiness to Change Drinking Behavior
Description: We will assess readiness to change with the Stages of Change Readiness and Treatment Eagerness Scale (SOCRATES), Version 8.This instrument was created by one of the initial developers of Motivational Interviewing, the therapeutic style on which SBIRT is based. SOCRATES is a 19-item instrument with 3 subscales where minimum score is 19 and the maximum score is 95. Lower totals representing lesser readiness/eagerness for change and higher totals representing greater readiness/eagerness to change. With the three sub scales (Recognition, Ambivalence, and Taking Steps), higher scores indicate greater recognition, ambivalence and taking steps and scores range from 7 to 35, 4 to 20, and 8 to 40, respectively.
Time Frame: 6 months
Population: Individuals that completed the 6 month interview
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Brief Alcohol Intervention (BI): 3-part Brief Intervention
  Brief Alcohol Intervention: 3 part intervention: Part I is 15-minute multi-component motivational discussion in hospital which includes personalized risk feedback, advice to abstain or reduce consumption, and the negotiation of an individual change plan. Part II is 15-minute follow-up in hospital to reinforce Part I. Part III is 15-minute follow-up telephone call at 2 weeks to reinforce Part I.
Arm/Group | Brief Alcohol Intervention (BI) | Attention Control | Control
Number analyzed (Participants) | 32 | 17 | 22
units on a scale | 23.16 (9.09) | 17.88 (8.48) | 17.00 (6.52)

5. Secondary Outcome: Adverse Consequences of Alcohol Use
Description: We will assess adverse consequences of alcohol use with the Short Inventory of Problems (SIP-2R), a widely used 15-item stand-alone short version of the Drinker Inventory of Consequences (DrInC).The SIP-2R will be administered at baseline (for BI and Attention Control) and at 6 months post-hospital discharge (all groups) to assesses adverse consequences of alcohol use over the past three months in five areas: Interpersonal, Physical, Social, Impulsive, and Intrapersonal. The SIP-2R was used as a continuous measure with possible scores from 0-45, where each item has a score from 0-3 (0=Never, 1=once or a few times, 2=once or twice a week, 3=daily or almost daily). Higher scores indicate a worse outcome.
Time Frame: 6 months
Population: Participants the completed the 6 month interview
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Brief Alcohol Intervention (BI) | Attention Control | Control
Number analyzed (Participants) | 32 | 17 | 22
units on a scale | 5.09 (3.03) | 5.41 (2.98) | 5.27 (2.35)

6. Other Pre Specified Outcome: Number of Participants Who Were Interested and Motivated to Change Their Alcohol Consumption
Description: Among Veterans randomized to Arm 1, we will analyze the transcripts of Part I of the audio-recorded brief intervention. Descriptive statistics (e.g., frequency distributions, measures of central tendency) will be used to characterize the anonymous sociodemographic, educational, and patient care characteristics of the participants. Transcript data will be analyzed using the grounded theory technique of constant comparison. Similar or related codes will be collapsed into focused codes in order to represent interrelationships, variations, and underlying patterns in the data, allowing for the identification of factors, issues, and themes related to Veterans interest and motivation for changing their alcohol consumption.
Time Frame: Baseline
Population: Data were not collected from the Attention Control and Control Groups
Measure: Count of Participants; unit: Participants
Groups:
- Brief Intervention: 3-part Brief Intervention. Part I is 15-minute multi-component motivational discussion in hospital which includes personalized risk feedback, advice to abstain or reduce consumption, and the negotiation of an individual change plan. Part II is 15-minute follow-up in hospital to reinforce Part I. Part III is 15-minute follow-up telephone call at 2 weeks to reinforce Part I.
  Brief Alcohol Intervention: 3 part intervention: Part I is 15-minute multi-component motivational discussion in hospital which includes personalized risk feedback, advice to abstain or reduce consumption, and the negotiation of an individual change plan. Part II is 15-minute follow-up in hospital to reinforce Part I. Part III is 15-minute follow-up telephone call at 2 weeks to reinforce Part I.
- Attention Control: Participants in this arm will complete all the screening and outcome measures that the Brief Intervention participants complete but will not receive any of the Brief Intervention treatments. They will receive a set of educational brochures/brochures which contain information and tips for healthy lifestyle behaviors such as alcohol and tobacco use, weight management, and physical activity to discuss with the Research Assistant. Approximately two weeks later, the Research Assistant will call patients in this condition at home for a 5-15 minute session to review the brochures and discuss any questions that s(he) may have.
  Lifestyle brochures: Set of educational brochures/brochures which contain information and tips for healthy lifestyle behaviors such as alcohol and tobacco use, weight management, and physical activity to discuss with the Research Assistant.
- Control: Participants in this arm will complete only drinking quantity measures at baseline and 6 months post baseline. They will receive a set of educational brochures/brochures which contain information and tips for healthy lifestyle behaviors such as alcohol and tobacco use, weight management, and physical activity to discuss with the Research Assistant. Approximately two weeks later, the Research Assistant will call patients in this condition at home for a 5-15 minute session to review the brochures and discuss any questions that s(he) may have.
  Lifestyle brochures: Set of educational brochures/brochures which contain information and tips for healthy lifestyle behaviors such as alcohol and tobacco use, weight management, and physical activity to discuss with the Research Assistant. Approximately two weeks later, the Research Assistant will call patients in this condition at home for a 5-15 minute session to review the brochures and discuss any questions that s(he) may have.
Arm/Group | Brief Intervention | Attention Control | Control
Number analyzed (Participants) | 37 | 0 | 0
Participants | 37 |  |

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Brief Alcohol Intervention (BI) | Attention Control | Control
All-Cause Mortality (participants affected / at risk) | 1/37 | 3/23 | 0/22
Serious Adverse Events (participants affected / at risk) | 0/37 | 0/23 | 0/22
Other Adverse Events (participants affected / at risk) | 5/37 | 0/23 | 0/22
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Brief Alcohol Intervention (BI) (N=37) | Attention Control (N=23) | Control (N=22)
Unable to administer part B of intervention (Investigations) | 3 | 0 | 0
Participant became alcohol dependent (Psychiatric disorders) | 1 | 0 | 0 — Participants in the study had to be hazardous drinkers -- after enrollment this participant became alcohol dependent
Participant entered palliative care (General disorders) | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes